CLINICAL TRIAL: NCT02930291
Title: The Effect of Preoperative Inflammation-based Scores on Postoperative Morbidity and Mortality for Laparoscopic Gastrectomy- A Prospective Cohort Study
Brief Title: The Effect of Preoperative Inflammation-based Scores on Postoperative Morbidity and Mortality for Laparoscopic Gastrectomy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Chang-Ming Huang, Prof., Director, Principal Investigator, Clinical Professor, Fujian Medical University
Other Study IDs: 2016YF017-02
Record Dates: First submitted 2016-09-21; First posted 2016-10-12 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Stomach Neoplasms
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to explore the effect of preoperative inflammation-based scores on postoperative morbidity and mortality for laparoscopic gastrectomy.

DETAILED DESCRIPTION:
A prospective cohort study will be performed to explore the effect of preoperative inflammation-based scores on postoperative morbidity and mortality for laparoscopic gastrectomy.The evaluation parameters are perioperative clinical efficacy, postoperative complications and 3-year survival and recurrence rates.

ELIGIBILITY:
Inclusion Criteria:Age from 18 to 75 years

* Primary lower third gastric adenocarcinoma (papillary, tubular, mucinous, signet ring cell, or poorly differentiated) confirmed pathologically by endoscopic biopsy
* cT2-4a, N0-3, M0 at preoperative evaluation according to the American Joint Committee on Cancer (AJCC) Cancer Staging Manual Seventh Edition
* No distant metastasis is observed. And the spleen, pancreas or other adjacent organs are not involved by the tumor.
* Performance status of 0 or 1 on Eastern Cooperative Oncology Group scale (ECOG)
* American Society of Anesthesiology score (ASA) class I, II, or III
* Written informed consent

Exclusion Criteria:• Women during pregnancy or breast-feeding

* Severe mental disorder
* History of previous upper abdominal surgery (except laparoscopic cholecystectomy)
* History of previous gastrectomy, endoscopic mucosal resection or endoscopic submucosal dissection
* Enlarged or bulky regional lymph node envelop important vessels
* History of other malignant disease within past five years
* History of previous neoadjuvant chemotherapy or radiotherapy
* History of unstable angina or myocardial infarction within past six months
* History of cerebrovascular accident within past six months
* History of continuous systematic administration of corticosteroids within one month
* Requirement of simultaneous surgery for other disease
* Emergency surgery due to complication (bleeding, obstruction or perforation) caused by gastric cancer
* FEV1<50% of predicted values

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who undergoing laparoscopic radical gastrectomy for gastric cancer are included.
Sampling Method: Non-Probability Sample
Enrollment: 310 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
3-year disease free survival rate | 36 months

SECONDARY OUTCOMES:
3-year disease overall survival rate | 36 months
Morbidity and mortality | 30 days; 36 months
  The early postoperative complication and mortality are defined as the event observed within 30 days after surgery, while the time frame for late complication is the period from postoperative day 31th to the end of month 36th.
3-year recurrence pattern | 36 months
Time to first ambulation | 10 days
  The data of postoperative recovery course.
The number of lymph node dissection | 1 day
The variation of weight | 12 months
  The variation of weight on postoperative 3, 6, 9 and 12 months
The daily highest body temperature | 7 day
  The daily highest body temperature before discharge
Time to first flatus | 10 days
Time to first liquid diet | 10 days
Time to soft diet | 10 days
Duration of hospital stay | 10 days
Intraoperative lymph node dissection time | 1 days
  intraoperative lymph node dissection time includes infrapyloric area lymph node,suprapancreatic area lymph
The amount of abdominal drainage | 10 days
Blood transfusion | 10 days
The number of positive lymph nodes | 1 day
Intraoperative morbidity rates | 1 day
  The intraoperative postoperative morbidity rates are defined as the rates of event observed within operation.
The rate of conversion to laparotomy | 1 day
The variation of cholesterol | 12 months
  The variation of cholesterol on postoperative 3, 6, 9 and 12 months
The variation of albumin | 12 months
  The variation of albumin on postoperative 3, 6, 9 and 12 months
The results of endoscopy | 12 months
  the results of endoscopy on postoperative 3 and 12 months
The values of white blood cell count | Preoperative 3 days and postoperative 1, 3, and 5 days
  The values of white blood cell count from peripheral blood before operation and on postoperative day 1, 3, 5 are recorded to access the inflammatory and immune response.
The values of lymphocyte count | Preoperative 3 days and postoperative 1, 3, and 5 days
  The values of lymphocyte count from peripheral blood before operation and on postoperative day 1, 3, 5 are recorded to access the inflammatory and immune response.
The values of neutrophil differential count | Preoperative 3 days and postoperative 1, 3, and 5 days
  The values of neutrophil differential count from peripheral blood before operation and on postoperative day 1, 3, 5 are recorded to access the inflammatory and immune response.
The values of platelet count | Preoperative 3 days and postoperative 1, 3, and 5 days
  The values of platelet count from peripheral blood before operation and on postoperative day 1, 3, 5 are recorded to access the inflammatory and immune response.
The values of hemoglobin | Preoperative 3 days and postoperative 1, 3, and 5 days
  The values of hemoglobin in gram/liter from peripheral blood before operation and on postoperative day 1, 3, 5 are recorded to access the inflammatory and immune response.
The values of C-reactive protein | Preoperative 3 days and postoperative 1, 3, and 5 days
  The values of C-reactive protein IN milligram/liter from peripheral blood before operation and on postoperative day 1, 3, 5 are recorded to access the inflammatory and immune response.
The values of prealbumin | Preoperative 3 days and postoperative 1, 3, and 5 days
  The values of prealbumin in gram/liter from peripheral blood before operation and on postoperative day 1, 3, 5 are recorded to access the inflammatory and immune response.
Visual Analog Score for pain | 7 days
  the values of visual analog score for pain before operation and on postoperative day 1 to day 7 are recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Changming Huang, Professor, Principal Investigator — Fujian Medical University Union Hospital,China
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No